CLINICAL TRIAL: NCT05670639
Title: CAPABLE Care Partner Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00308713
Record Dates: First submitted 2022-12-13; First posted 2023-01-04 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Aging; Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot (Other)
  Interventions: Behavioral: CAPABLE Care Partner

INTERVENTIONS:
Behavioral: CAPABLE Care Partner — The CAPABLE Care Partner intervention consists of three components: 1) up to 3 sessions with a Care Partner Support person focused on developing action plans for self-care goals of the care partner 2) educational materials provided in a folder at the beginning of the program 3) inclusion in the CAPABLE clinician visits as deemed appropriate by the client, CAPABLE clinicians, and care partner

SUMMARY:
This is a small-scale multi-site pilot of a supplemental enhancement called "Care Partner" to the evidence-based CAPABLE program that will involve up to 60 individuals (30 care partners and older adult dyads) and 30 professional staff in organizations currently licensed to provide CAPABLE. This is a qualitative study of a convenience sample of individuals.

DETAILED DESCRIPTION:
Care partners (family/friend caregivers) of older adults are integral to the ability of these individuals to remain living in the community as independently as possible. Through the 12-year history of developing and offering CAPABLE, particularly the last four years when the program has been nationally disseminated, CAPABLE sites across the country have observed that in about 25% of cases, the older adult participant has a family or friend care partner who either lives with the older person (usually a spouse/partner) or is significantly involved in providing care or support with activities of daily living. This is consistent with other research on the level of caregiving in the U.S which indicates from 21-25% of individuals in the U.S. provided care to a family member or friend with a health limitation or disability within the last 30 days.

The evidence-based CAPABLE program developed by Drs. Gitlin and Szanton of Johns Hopkins School of Nursing does not currently have a structured or consistent way to involve these care partners in CAPABLE, nor does it offer any support to the care partner directly. Research on caregivers indicates that from 20-50% report delaying or skipping care as a result of focusing on caregiving for others and that caregiving has negatively impacted the caregivers own health status. However, there are positive aspects of caregiving as well, including deepening the relationship and enhancing the sense of purpose for the caregiver. The Centers for Disease Control and Prevention have identified need for support to caregivers in the Public Health Call to Action.

In Phases 1 and 2 of this CAPABLE Care Partner study (completed), the investigators co-created the Care Partner component as an add-on to CAPABLE, working with caregiving experts, CAPABLE clinicians, older adults, and care partners.

The purpose of this Care Partner Pilot Study is to:

1. develop a prototype for an enhanced component to CAPABLE, focusing on the family or friend caregiver (called Care Partner) and
2. evaluate the prototype through a multi-site pilot so it can be used by existing sites.

This pilot focuses on feasibility and acceptability of the Care Partner component, and a preliminary assessment of the effect on care partners.

The objectives are:

* Assess the feasibility of the CAPABLE Care Partner component being integrated into CAPABLE from the perspective of CAPABLE participants, care partners, CAPABLE program administrators, CAPABLE clinicians, and the Care Partner Support Specialist
* Determine the acceptability of CAPABLE Care Partner component to CAPABLE participants, care partners, CAPABLE program administrators, CAPABLE clinicians, and the Care Partner Support Specialist
* Evaluate effect of the Care Partner component on care partners, measuring self-reported competency, well-being, and indicators of stress, and obtaining qualitative information from a convenience sample of care partners.

ELIGIBILITY:
Inclusion Criteria:

Care Partner:

* Provides 10+ hours/week of care or support for CAPABLE program participant
* Able to participate in two 45 minutes phone interview or virtual meetings
* English-speaking

CAPABLE Participant:

* CAPABLE participant of one of the CAPABLE programs offered by a pilot site organization
* Able to participate in two 30-minute phone interview or virtual meetings
* English-speaking

Occupational Therapist (OT)/ Registered Nurse (RN):

* Has been trained to provide CAPABLE and has served CAPABLE clients for at least 6 months
* Currently serving CAPABLE participants
* Able to participate in two one-hour phone call or virtual meetings
* English-speaking

Care Partner Support Specialist

* Licensed social worker or other professional trained in providing caregiver support
* Able to participate in two one-hour phone call or virtual meetings
* English-speaking

Program Administrator

* Currently managing a CAPABLE program
* Able to participate in two one-hour phone call or virtual meetings
* English-speaking

Exclusion Criteria: Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Level of acceptance of intervention as assessed by qualitative assessments | 10-12 months
  Qualitative interviews with each type of key informant at the end of the pilot will help us understand the level of acceptance of the Care Partner addition by each subject type (i.e., care partner, clinician, administrator). An adjectival scale will be used with 4 points from "Very satisfied to Very unsatisfied" together with open-ended questions.
Potential barriers and catalysts in implementation as assessed by key informant interviews with program administrators via semi-structured interview guide | 10 months
  Potential barriers and catalysts in implementation for incorporating Care Partners into CAPABLE-including the feasibility related to costs, resources, and other factors through key informant interviews with the program administrators using a semi-structured interview guide. An Adjectival scale will be used with 4 points from "Very satisfied to Very unsatisfied" together with open-ended questions.
Change in Depression as assessed by the Patient Health Questionnaire Depression Scale (PHQ-2) | Baseline, 4 months - at the end of the intervention for each care partner
  The PHQ-2 screening instrument contains 2 questions, 4-point Adjectival Likert scale from "Not at all" to "Nearly every day" with the "nearly every day" response indicating more severe depressive symptoms.
Change in self-reported health status as assessed by one item in the 12-item Short Form Survey (SF-12) | Baseline, 4 months at the completion of the intervention for each care partner
  The SF-12 is a 12-item questionnaire with a 5-point Likert scale (responses ranging from 'excellent' to 'poor'). The self-report of "fair" or "poor" indicates worse self-reported health status and has shown predictive power associated with higher morbidity or mortality.
Change in the perception of caregiving effectiveness as measured by the Caregiving Effectiveness Scale (Noelker) | Baseline, 4 months at the completion of the intervention for each care partner
  Two items from the Caregiving Effectiveness scale with a 4-point adjectival Likert scale (responses ranging from 'very satisfied' to 'not satisfied at all'. A response of "not satisfied at all" indicates lower perception of caregiving effectiveness.
Change in caregiving competence and confidence as assessed by the Pearlin's Caregiving Competence Scale. | Baseline, 4 months at completion of the intervention for each care partner
  Two items using a 5-point adjectival Likert scale (responses ranging from "Strongly disagree to Strongly Agree). A higher score (agreement) would indicate higher competency/satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No